CLINICAL TRIAL: NCT00642889
Title: A PHASE III, DOUBLE-BLIND, PLACEBO-CONTROLLED, 12-MONTH EXTENSION STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF A DOSE RANGE OF SAFINAMIDE OF 50-200 MG/DAY, AS ADD-ON THERAPY IN PATIENTS WITH EARLY IDIOPATHIC PARKINSON'S DISEASE TREATED WITH A STABLE DOSE OF A SINGLE DOPAMINE AGONIST.
Brief Title: Safinamide as Add-On Therapy in Patients With Early Idiopathic Parkinson's Disease Treated With a Stable Dose of a Single Dopamine Agonist (12 Month Extension)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Dr Stefano Rossetti, Newron Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW-1015/017/III/2003
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Dose (Experimental): 150-200mg/day
  Interventions: Drug: Safinamide
- Low dose (Experimental): 50-100mg/day
  Interventions: Drug: Safinamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Safinamide
  Arms: High Dose
Drug: Safinamide
  Arms: Low dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
To determine the long-term safety and efficacy of a dose range of safinamide of 50-200 mg/day, p.o., compared to placebo, as add-on therapy in patients with early idiopathic Parkinson's disease who are currently receiving a stable dose of a single dopamine (DA) agonist.

DETAILED DESCRIPTION:
The study will consist of 12 months of double-blind treatment. Patients will continue to take the original treatment administered in Study 015 (safinamide 100 mg/day, safinamide 200 mg/day, or placebo).

ELIGIBILITY:
Inclusion Criteria:

1. The patient completed 24 weeks of treatment in Study 015, or if the patient discontinued prematurely, he/she returned for scheduled efficacy evaluations at Weeks 12 and 24 (Visits 6 and 8) as part of the Retrieved Dropout (RDO) population.
2. The patient was compliant with taking study medication in Study 015.
3. The patient is willing to participate in the study and signed an approved Informed Consent form.

Exclusion Criteria:

1. The patient is experiencing clinically significant adverse events that would put the patient at risk for participating in the study.
2. The patient has shown clinically significant deterioration during participation in Study 015.
3. The patient discontinued Study 015 prematurely for any reason, and did not return for scheduled efficacy evaluations at Weeks 12 and 24 (Visits 6 and 8) in Study 015.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2005-06; Primary Completion 2007-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time from baseline to intervention (e.g., increase in dose of DA-agonist; addition of another DA-agonist, levodopa, or other PD therapy; or discontinuation due to lack of efficacy); or time from baseline to the last follow up, if the event did not occur